CLINICAL TRIAL: NCT04887402
Title: Different Variables Predicting Ovulatory Response Among Clomiphene Citrate Resistance and Clomiphene Citrate Sensitive Patients With Polycystic Ovarian Syndrome.
Brief Title: Parameters Declaring PCO Infertile Patients Either Sensitive or Resistant to Different Doses of Clomiphene Citrate.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Alaa Sherif Zakaria Saad Elsewafy, Assistant lecturer, Ain Shams Maternity Hospital
Other Study IDs: Parameters of resistence
Record Dates: First submitted 2021-05-11; First posted 2021-05-14 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: PCO; Induction of Ovulation; Clomiphene Citrate
Keywords: induction of ovulation by clomiphene citrate in PCO
MeSH Terms: interventions — Clomiphene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- clomiphene citrate sensitive: Based on the ovulation pattern, these patients will be divided into two groups, one who ovulated with CC maximum 150 mg and others who did not ovulate considered as CC resistant. The patients who ovulated will be further classified into three subgroups based on whether they ovulated with 50 mg or 100 mg or 150 mg of CC.
  The various parameters will be compared between the CC-resistant and CC-sensitive groups.
  Interventions: Drug: Clomiphene Citrate
- clomiphene citrate resistent: Based on the ovulation pattern, these patients will be divided into two groups, one who ovulated with CC maximum 150 mg and others who did not ovulate considered as CC resistant. The patients who ovulated will be further classified into three subgroups based on whether they ovulated with 50 mg or 100 mg or 150 mg of CC.
  The various parameters will be compared between the CC-resistant and CC-sensitive groups.
  Interventions: Drug: Clomiphene Citrate

INTERVENTIONS:
Drug: Clomiphene Citrate — All patients will be treated with CC starting with 50 mg/day on the day 2 of their cycle for 5 days, a transvaginal ultrasound will be done 1 week after the last pill, if all follicles are below 10 mm the dose will subsequently be increased to 100mg/day for 5 days then 150mg/day for 5 days if a transvaginal is done a week from the last pill and showed no response (all follicles being below 10 mm ).Maximum cc dose will be 150 mg (ASRM, 2013). Medroxyprogesterone (10 mg/d Provera for 10 days)will be given to induce withdrawal bleeding to start these steps again in a new cycle. These steps will be repeated for 3cycles before declaring the patient CC resistant.
  o Response: Response to CC will be assessed by ovulation. TVS will be done by the same observer using a Samsung ultrasound machine, HS40.
  A scan will be done 1 week after the last pill of each dose. No response: if all follicles are below 10 mm (ASRM, 2013), follicles >10mm, follow up till ovulation

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common endocrinological disorder seen in 6%-10% of women (Human Reproduction, 2004). It is characterized by polycystic ovaries, anovulatory cycles, and hyperandrogenism.

In nearly 20% of infertile women, PCOS is said to be the key reason behind infertility (Norman et al., 2007).

PCOS is a syndrome that manifests variably from adolescence as oligomenorrhea or hirsutism or obesity and goes on to affect the reproductive performance of the female by causing anovulation. Some may even be severely affected by metabolic syndrome, diabetes mellitus, or endometrial carcinoma. It also increases the risk of ovarian and breast carcinoma (Atiomo et al., 2003).

PCOS falls in WHO type II anovulation (norm-gonadotropic norm-estrogenic anovulation) and is seen in 85% of anovulatory females. Although lifestyle modification is known to improve reproductive outcomes in females with PCOS, the gold standard treatment for norm-gonadotropic oligo/amenorrheic infertility (WHO Group II) was clomiphene citrate (CC) (Radosh L., 2009) until 2018, when ESHRE and ASRM have declared letrozole as the first-line treatment for ovulation induction (OI)( ESHRE 2018 guidelines).

To conclude, available data shows that letrozole is at least as effective as CC for ovulation and has comparable live birth rates. Importantly, it has definite advantages over CC. Many studies have shown letrozole to be as effective as gonadotropins, with added advantage of low cost and lower multiple pregnancy rates. However, the quality of medical evidence supporting aromatase inhibitors for OI, are inadequate, small in sample size, and inappropriate design. Moreover, there is very limited data on potential teratogenic effects, oocyte, embryo quality, and any effect on implantation. ( Misso et al., 2012) Those who fail to respond to CC are labeled as clomiphene resistant. It is common in approximately 15%-40% of women with PCOS (NICE, 2014). Major factors postulated for CC resistance include obesity, insulin resistance, (seen in nearly 50%-70% of females with PCOS) and hyperandrogenemia (Parsanezhad et al., 2001).Moreover, genetic predisposition is suggested to play a role in CC resistance (Overbeek et al., 2009).However, still, the current data available on the causes of CC resistance are not sufficient enough to direct our treatment.

It is seen in various studies (Sohrevardi et al.,2016) that the females who initially failed to respond to CC develop better ovulation and pregnancy outcomes on treatment with insulin-sensitizing agents. This indicates that insulin resistance may be a cause of CC resistance in females with PCOS. In fact, insulin-sensitizing agents (Azziz et al., 2009) decrease the dose of ovulation-inducing agent and time for follicular maturation in females with PCOS.

As of now, there have been no concrete studies to compare the metabolic profile of females who respond to CC and those who do not. It is still an enigma as to why some women respond to clomiphene, while others do not. By identifying the various factors which affect the response of CC in patients with infertility, a lot of time can be saved by giving alternate options of treatment to these patients. This study was done with the aim to analyze various clinical, metabolic, hormonal, and ultrasound parameters that might affect the response to clomiphene.

DETAILED DESCRIPTION:
All PCO patients under the age of 40 who are subfertile with no identified cause but PCO will undergo the following;

* Detailed history taking including age, parity, medical, surgical history, previous trials of induction of ovulation.
* Physical examination:

  * Vital data: blood pressure
  * General examination: including weight in kilograms, and height in an upright posture without shoes using to the nearest 0.5 cm will be recorded. Body mass index (BMI) will be recorded from the above measurements. Waist circumference (WC) will be measured midway between the lower rib margin and the iliac crest in the mid-axillary line at the end of normal expiration. Hip circumference will be measured with the measuring tape at the highest prominence of the buttocks and parallel to the floor (Nishida et al., 2010). WC and hip circumference will be recorded after removing clothing from the area over the waist and hip.

The thyroid will be examined for any enlargement, nodules, or tenderness. The breast will be examined for any enlargement or galactorrhea. Signs of androgen excess will be looked for such as; excessive hair growth, acne, or alopecia. Excessive hair growth will be evaluated by modified Ferriman and Gallwey (Wild et al., 2004) (FG) score(<8 normal,8-15mild hirsutism,>15 moderate/severe hirsutism).

* Abdominal examination: including the presence of previous scars, uterine size, any tenderness, and presence of palpable masses, score on Ferriman Gallway scoring system.
* Pelvic examination: including uterine size, any adnexal mass, and tenderness, score on Ferriman Gallway scoring system.

  o Investigation:

  a) Laboratory (on the 2nd day of cycle):
* Serum testosterone
* Androstenedione
* AMH
* LH
* FSH
* Fasting and 2hrs postprandial b) Imaging -Transvaginal ultrasound(on the 2nd day of cycle):
* Antral follicular count (AFC)
* Ovarian volume
* Endometrial thickness Will be done by the same observer using a Samsung ultrasound machine, HS40 (TVS probe frequency range 5-7 MHZ). The ovarian volume of each ovary will be assessed by ellipsoid formula, i.e., 0.52 × D1 (longitudinal) × D2 (oblique) × D3 (transverse) diameters. Mean ovarian volume will be calculated by adding the volume of both ovaries and then dividing it by 2. A note of ovarian follicles in each ovary will be also made and a total number of the follicles will be counted by scanning each ovary from the inner to the outer margin in longitudinal cross-section. Mean follicle number will be calculated by adding the follicles of both ovaries and then dividing it by 2.

  * Method (stair step protocol):

All patients will be treated with CC starting with 50 mg/day on day 2 of their cycle for 5 days, a transvaginal ultrasound will be done 1 week after the last pill, if all follicles are below 10 mm the dose will subsequently be increased to 100mg/day for 5 days then 150mg/day for 5 days if a transvaginal is done a week from the last pill and showed no response (all follicles being below 10 mm ). The maximum cc dose will be 150 mg (ASRM, 2013). Medroxyprogesterone (10 mg/d Provera for 10 days)will be given to induce withdrawal bleeding to start these steps again in a new cycle. These steps will be repeated for 3cycles before declaring the patient CC resistant.

o Response: Response to CC will be assessed by ovulation. TVS will be done by the same observer using a Samsung ultrasound machine, HS40.

A scan will be done 1 week after the last pill of each dose. No response: if all follicles are below 10 mm (ASRM, 2013), follicles >10mm, follow up till ovulation Based on the ovulation pattern, these patients will be divided into two groups, one who ovulated with CC maximum 150 mg and others who did not ovulate considered as CC resistant. The patients who ovulated will be further classified into three subgroups based on whether they ovulated with 50 mg or 100 mg or 150 mg of CC.

The various parameters will be compared between the CC-resistant and CC-sensitive groups.

ELIGIBILITY:
Inclusion Criteria:

* PCOS (based on Rotterdam's criteria: oligo/anovulation, hyperandrogenism clinical (hirsutism or less commonly male pattern alopecia) /biochemical (raised FAI or free testosterone) or polycystic ovaries on ultrasound(presence of 12 or more follicles in each ovary measuring 2-9 mm in diameter, and/or increased ovarian volume (>10 ml)"1 . Unilaterality does not affect diagnosis; neither does the location of the cysts in the ovary.)
* Age <40 years.
* Semen analysis within normal according to WHO 2010.

Exclusion Criteria:

* Women on any insulin-sensitizing agent.
* Women on lipid-lowering agent.
* Women with endocrinal disorder (such as thyroid dysfunction, insulin resistance(DM), and adrenal disorders).
* Women diagnosed with anorexia nervosa/bulimia nervosa.
* Women with hypothalamic or pituitary dysfunction.
* Age >40
* AMH level that does not reflect the phenotype of PCO

Max Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will include 100 women with PCO Using PASS 11 program for sample size calculation and according to (sachdeva etal,2019), the expected frequency of PCOs patients with CC resistance = 54%, assuming that frequency in study population =54%+\- 10% and at 95% confidence level, sample size of 100 patients will be enough to detect this frequency.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
ovulation | maximum 3 months
  follow up patient response to induction of ovulation by folliculometry till ovulation occurs

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Rateb, professor, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Atiomo WU, El-Mahdi E, Hardiman P. Familial associations in women with polycystic ovary syndrome. Fertil Steril. 2003 Jul;80(1):143-5. doi: 10.1016/s0015-0282(03)00502-8. PMID 12849816
- [Result] Azziz R, Carmina E, Dewailly D, Diamanti-Kandarakis E, Escobar-Morreale HF, Futterweit W, Janssen OE, Legro RS, Norman RJ, Taylor AE, Witchel SF; Task Force on the Phenotype of the Polycystic Ovary Syndrome of The Androgen Excess and PCOS Society. The Androgen Excess and PCOS Society criteria for the polycystic ovary syndrome: the complete task force report. Fertil Steril. 2009 Feb;91(2):456-88. doi: 10.1016/j.fertnstert.2008.06.035. Epub 2008 Oct 23. PMID 18950759
- [Result] Misso ML, Wong JL, Teede HJ, Hart R, Rombauts L, Melder AM, Norman RJ, Costello MF. Aromatase inhibitors for PCOS: a systematic review and meta-analysis. Hum Reprod Update. 2012 May-Jun;18(3):301-12. doi: 10.1093/humupd/dms003. Epub 2012 Mar 19. PMID 22431566
- [Result] Norman RJ, Dewailly D, Legro RS, Hickey TE. Polycystic ovary syndrome. Lancet. 2007 Aug 25;370(9588):685-97. doi: 10.1016/S0140-6736(07)61345-2. PMID 17720020
- [Result] Overbeek A, Kuijper EA, Hendriks ML, Blankenstein MA, Ketel IJ, Twisk JW, Hompes PG, Homburg R, Lambalk CB. Clomiphene citrate resistance in relation to follicle-stimulating hormone receptor Ser680Ser-polymorphism in polycystic ovary syndrome. Hum Reprod. 2009 Aug;24(8):2007-13. doi: 10.1093/humrep/dep114. Epub 2009 Apr 28. PMID 19401323
- [Result] Parsanezhad ME, Alborzi S, Zarei A, Dehbashi S, Omrani G. Insulin resistance in clomiphene responders and non-responders with polycystic ovarian disease and therapeutic effects of metformin. Int J Gynaecol Obstet. 2001 Oct;75(1):43-50. doi: 10.1016/s0020-7292(01)00470-2. PMID 11597618
- [Result] Radosh L. Drug treatments for polycystic ovary syndrome. Am Fam Physician. 2009 Apr 15;79(8):671-6. PMID 19405411
- [Result] Dunaif A, Fauser BC. Renaming PCOS--a two-state solution. J Clin Endocrinol Metab. 2013 Nov;98(11):4325-8. doi: 10.1210/jc.2013-2040. Epub 2013 Sep 5. PMID 24009134
- [Result] Sohrevardi SM, Nosouhi F, Hossein Khalilzade S, Kafaie P, Karimi-Zarchi M, Halvaei I, Mohsenzadeh M. Evaluating the effect of insulin sensitizers metformin and pioglitazone alone and in combination on women with polycystic ovary syndrome: An RCT. Int J Reprod Biomed. 2016 Dec;14(12):743-754. PMID 28331909
- [Result] WHO Expert Consultation. Appropriate body-mass index for Asian populations and its implications for policy and intervention strategies. Lancet. 2004 Jan 10;363(9403):157-63. doi: 10.1016/S0140-6736(03)15268-3. PMID 14726171
- [Result] 11. Wild, R.A., 2004. Ferriman Gallwey self-scoring: Performance assessment in women with the polycystic ovary syndrome (Doctoral dissertation, The University of Oklahoma Health Sciences Center).
- [Result] Practice Committee of the American Society for Reproductive Medicine. Use of clomiphene citrate in infertile women: a committee opinion. Fertil Steril. 2013 Aug;100(2):341-8. doi: 10.1016/j.fertnstert.2013.05.033. Epub 2013 Jun 27. PMID 23809505